CLINICAL TRIAL: NCT00767806
Title: Effect of Duloxetine 60 mg Once Daily Versus Placebo in Patients With Chronic Low Back Pain
Brief Title: A Study for Patient With Chronic Low Back Pain
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Chief Medical Officer, Eli Lilly
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 12360; F1J-MC-HMGC (Other: Eli Lilly and Company)
Record Dates: First submitted 2008-10-03; First posted 2008-10-07 (Estimated); Results first posted 2010-10-18 (Estimated); Last update posted 2010-10-18 (Estimated); Status verified 2010-09

CONDITIONS: Chronic Low Back Pain
MeSH Terms: interventions — Duloxetine Hydrochloride

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Duloxetine (Experimental): Participants received duloxetine 60 milligram by mouth once daily for 12 weeks of double-blind treatment
  Interventions: Drug: Duloxetine
- Placebo (Placebo Comparator): Patients received placebo by mouth once daily for 12 weeks of double-blind treatment
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Duloxetine — 60 mg orally once daily for 12 weeks
  Other Names: Cymbalta; LY248686
  Arms: Duloxetine
Drug: Placebo — Placebo once daily orally for 12 weeks
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine if duloxetine reduces the severity of chronic low back pain.

ELIGIBILITY:
Inclusion Criteria:

* Male or female outpatients with chronic low back pain

Exclusion Criteria:

* Cardiovascular, hepatic, renal, respiratory, or hematologic illness, or other medical or psychiatric condition that, in the opinion of the investigator, would compromise participation or be likely to lead to hospitalization during the course of the study.
* Acute liver injury (such as hepatitis) or severe cirrhosis.
* Previous exposure to duloxetine.
* Body Mass Index (BMI) over 40.
* Major depressive disorder.
* Daily use of narcotics.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 401 (Actual)
Dates: Start 2008-09; Primary Completion 2009-07 (Actual); Study Completion 2009-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559) or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (26):
- United States (7):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Chandler, Arizona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Cromwell, Connecticut
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., DeLand, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Jacksonville, Florida
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Brighton, Massachusetts
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Oklahoma City, Oklahoma
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Portland, Oregon
- Brazil (2):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Sacomã
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., São Paulo
- Germany (6):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Aalen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Alzenau in Unterfranken
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Berlin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Ellwangen
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Hamburg
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Wiesbaden
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Rotterdam, Netherlands
- Poland (4):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Krakow
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Lublin
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Poznan
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Szczecin
- For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Moscow, Russia
- Spain (5):
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., A Coruña
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Barcelona
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Bilboa
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Getafe
  - For additional information regarding investigative sites for this trial, contact 1-877-CTLILLY (1-877-285-4559, 1-317-615-4559) Mon - Fri from 9 AM to 5 PM Eastern Time (UTC/GMT - 5 hours, EST), or speak with your personal physician., Madrid

REFERENCES:
- [Background] Skljarevski V, Zhang S, Desaiah D, Alaka KJ, Palacios S, Miazgowski T, Patrick K. Duloxetine versus placebo in patients with chronic low back pain: a 12-week, fixed-dose, randomized, double-blind trial. J Pain. 2010 Dec;11(12):1282-90. doi: 10.1016/j.jpain.2010.03.002. Epub 2010 May 15. PMID 20472510
- [Derived] Williamson OD, Schroer M, Ruff DD, Ahl J, Margherita A, Sagman D, Wohlreich MM. Onset of response with duloxetine treatment in patients with osteoarthritis knee pain and chronic low back pain: a post hoc analysis of placebo-controlled trials. Clin Ther. 2014 Apr 1;36(4):544-51. doi: 10.1016/j.clinthera.2014.02.009. Epub 2014 Mar 17. PMID 24650448

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Duloxetine | Placebo
Started | 198 | 203
Completed | 147 | 156
Not Completed | 51 | 47
Not completed — Adverse Event | 30 | 11
Not completed — Withdrawal by Subject | 8 | 13
Not completed — Protocol Violation | 6 | 5
Not completed — Lack of Efficacy | 1 | 9
Not completed — Physician Decision | 4 | 3
Not completed — Lost to Follow-up | 1 | 4
Not completed — Entry Criteria Not Met | 1 | 1
Not completed — Sponsor Decision | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Duloxetine | Placebo | Total
Number analyzed (Participants) | 198 | 203 | 401
Age Continuous [Mean (Standard Deviation); unit: years] | 54.87 (13.27) | 53.43 (14.17) | 54.14 (13.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 118 | 128 | 246
  Male | 80 | 75 | 155
Race/Ethnicity, Customized [Number; unit: participants]
  African | 5 | 5 | 10
  Caucasian | 189 | 193 | 382
  Hispanic | 4 | 4 | 8
  Native American | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 64 | 67 | 131
  Poland | 35 | 35 | 70
  Spain | 25 | 26 | 51
  Russian Federation | 35 | 33 | 68
  Netherlands | 16 | 16 | 32
  Germany | 23 | 26 | 49
Quebec Task Force on Spinal Disorders [Number; unit: participants] — Quebec Task Force: class 1: pain; class 2: pain with radiation to lower limb proximally. Data was not available for all participants.
  participants
    Class 1 | 173 | 168 | 341
    Class 2 | 21 | 30 | 51
    Not Available | 4 | 5 | 9
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram/meter squared] — The BMI is the weight of the participant divided by the squared height of the participant.
  kilogram/meter squared | 27.56 (4.50) | 28.14 (4.72) | 27.85 (4.62)
Brief Pain Inventory Average Pain Rating [Mean (Standard Deviation); unit: units on a scale] — A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine).
  units on a scale | 5.84 (1.43) | 5.75 (1.37) | 5.79 (1.40)
Clinical Global Impression - Severity (CGI-S) [Mean (Standard Deviation); unit: units on a scale] — CGI-S at baseline measures severity of illness at the start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients).
  units on a scale | 3.49 (1.24) | 3.29 (1.28) | 3.39 (1.27)
Duration of Chronic Lower Back Pain [Mean (Standard Deviation); unit: years] | 8.28 (8.18) | 8.74 (8.95) | 8.51 (8.57)
Height [Mean (Standard Deviation); unit: centimeter] | 168.24 (9.64) | 167.91 (8.82) | 168.07 (9.22)
Roland Morris Disability Questionnaire [Mean (Standard Deviation); unit: units on a scale] — Roland-Morris questionnaire will be completed by the patient and measures the degree of disability due to back pain. The questionnaire consists of 24 statements and the patient is instructed to put a mark next to each appropriate statement. The number of statements marked will be added up by the clinician and a total score is given. The total score ranges from 0 (no disability) to 24 (severe disability).
  units on a scale | 9.63 (4.64) | 9.32 (4.77) | 9.47 (4.70)
Weekly mean of 24-hour average pain rating using an 11-point numerical scale patient diary [Mean (Standard Deviation); unit: units on a scale] — 24-hour average pain severity scores recorded daily on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). Patients should complete the electronic diary at bedtime. The 11-point Likert scale will also be used for assessment of night pain and worst pain each day, and evaluated as weekly means.
  units on a scale | 5.79 (1.36) | 5.80 (1.37) | 5.80 (1.36)
Weight [Mean (Standard Deviation); unit: kilogram] | 78.30 (15.83) | 79.35 (14.65) | 78.83 (15.23)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to 12 Weeks in Brief Pain Inventory 24-hour Average Pain Score
Description: A self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Least Squares Mean values were controlled for investigator and baseline severity.
Time Frame: baseline, 12 weeks
Population: All randomized participants with baseline and at least 1 non-missing post-baseline value.
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 195 | 199
units on a scale | -2.48 (0.16) | -1.80 (0.15)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory 24-hour average pain score after 12 weeks of treatment; Test type: Superiority or Other; p = 0.001, Mixed Models Analysis

2. Secondary Outcome: Change From Baseline to 12 Weeks on the Brief Pain Inventory - Severity (BPI-S) and Interference (BPI-I)
Description: BPI-S and BPI-I are self-reported scales measuring severity of pain and interference on function. Severity scores: 0 (no pain) to 10 (severe pain) on each question assessing worst pain, least pain in past 24 hours, and pain right now. Interference scores: 0 (does not interfere) to 10 (completely interferes) on each question assessing interference of pain in past 24 hours for general activity, mood, walking ability, normal work, relations with other people, sleep, and enjoyment of life. Average interference = average of non-missing scores of individual interference items.
Time Frame: baseline, 12 weeks
Population: All randomized participants with baseline and at least 1 non-missing post-baseline value. Last observation carried forward method was used to impute missing endpoints.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 195 | 199
units on a scale
  BPI severity of worst pain - baseline | 7.26 (1.52) | 7.06 (1.54)
  BPI severity of worst pain - change | -2.75 (2.33) | -1.99 (2.29)
  BPI severity of least pain - baseline | 4.11 (2.07) | 4.04 (2.03)
  BPI severity of least pain - change | -1.67 (2.01) | -1.16 (2.04)
  BPI severity of pain right now - baseline | 5.47 (2.00) | 5.30 (1.84)
  BPI severity of pain right now - change | -2.55 (2.27) | -1.65 (2.05)
  BPI interference with general activity - baseline | 5.37 (2.33) | 4.91 (2.16)
  BPI interference with general activity - change | -2.71 (2.39) | -1.71 (2.30)
  BPI interference with mood - baseline | 4.00 (2.70) | 3.76 (2.54)
  BPI interference with mood - change | -2.26 (2.45) | -1.41 (2.40)
  BPI interference with walking ability - baseline | 4.61 (2.66) | 4.13 (2.57)
  BPI interference with walking ability - change | -2.23 (2.42) | -1.52 (2.27)
  BPI interference with normal work - baseline | 5.25 (2.33) | 4.91 (2.33)
  BPI interference with normal work - change | -2.50 (2.44) | -1.82 (2.22)
  BPI interference relations with others - baseline | 3.07 (2.67) | 2.82 (2.58)
  BPI interference relations with others - change | -1.74 (2.35) | -1.04 (2.37)
  BPI interference with sleep - baseline | 4.74 (2.89) | 4.53 (2.79)
  BPI interference with sleep - change | -2.37 (2.67) | -1.55 (2.55)
  BPI interference with enjoyment of life - baseline | 4.25 (2.84) | 3.78 (2.70)
  BPI interference with enjoyment of life - change | -2.44 (2.56) | -1.59 (2.55)
  BPI average interference - baseline | 4.44 (2.15) | 4.14 (2.08)
  BPI average interference - change | -2.26 (1.96) | -1.55 (1.93)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory severity of worst pain score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value is for BPI severity of worst pain - change; Main effect model: Change = Treatment + Investigator + Baseline (Type III sums of square); Mean Difference (Final Values) = -0.68, 95% CI 2-sided [-1.12 to -0.25]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory severity of least pain score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.006, ANCOVA — P-value is for BPI severity of least pain - change; Main effect model: Change = Treatment + Investigator + Baseline (Type III sums of square); Mean Difference (Final Values) = -0.49, 95% CI 2-sided [-0.85 to -0.14]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory severity of pain right now score during 12 weeks of treatment; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for BPI severity of pain right now - change; Main effect model: Change = Treatment + Investigator + Baseline (Type III sums of square); Mean Difference (Final Values) = -0.86, 95% CI 2-sided [-1.25 to -0.46]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory interference with general activity score during 12 weeks of treatment; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for BPI interference with general activity - change; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.75, 95% CI 2-sided [-1.16 to -0.35]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory interference with mood score during 12 weeks of treatment; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for BPI interference with mood score - change; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.09 to -0.34]
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory interference with walking ability score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.020, ANCOVA — P-value is for BPI interference with walking ability - change; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.46, 95% CI 2-sided [-0.84 to -0.07]
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory interference with normal work score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.012, ANCOVA — P-value is for BPI interference with normal work - change; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.51, 95% CI 2-sided [-0.90 to -0.11]
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory interference with relations to others score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.001, ANCOVA — P-value is for BPI interference with relations to others - change; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.92 to -0.22]
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory interference with sleep score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.002, ANCOVA — P-value is for BPI interference with sleep score - change; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.13 to -0.27]
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory interference with enjoyment of life score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.005, ANCOVA — P-value is for BPI interference with enjoyment of life score - change; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.96 to -0.18]
Statistical Analysis 11: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Brief Pain Inventory average interference score during 12 weeks of treatment; Test type: Superiority or Other; p < 0.001, ANCOVA — P-value is for BPI average interference score - change; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.58, 95% CI 2-sided [-0.92 to -0.25]

3. Secondary Outcome: Change From Baseline to 12 Weeks in Weekly Mean of 24-hour Average Pain, Worst Pain, and Night Pain Rating
Description: 24-hour average pain severity scores were recorded daily on an 11-point Likert scale, an ordinal scale ranging from 0 (no pain) to 10 (worst possible pain). Patients completed the electronic diary at bedtime. The 11-point Likert scale was also used for assessment of night pain and worst pain each day, and evaluated as weekly means. Least Squares Mean values were controlled for investigator and baseline severity.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 152 | 162
units on a scale
  Average Pain | -2.14 (0.14) | -1.43 (0.13)
  Worst Pain | -2.19 (0.15) | -1.48 (0.14)
  Night Pain | -1.62 (0.14) | -1.10 (0.14)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the weekly 24-hour average pain rating score during 12 weeks of treatment; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for weekly 24-hour average pain rating score - change; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.70, 95% CI 2-sided [-1.05 to -0.35]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the weekly 24-hour worst pain score during 12 weeks of treatment; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for weekly 24-hour worst pain score - change; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.71, 95% CI 2-sided [-1.08 to -0.33]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the weekly 24-hour night pain score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.004, ANCOVA — p-value is for weekly 24-hour night pain score - change; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.52, 95% CI 2-sided [-0.87 to -0.17]

4. Secondary Outcome: Number of Responders: 30 Percent (%) or Greater Reduction of the Brief Pain Inventory (BPI) Average Pain Severity Rating at 12 Week Endpoint
Description: Response to treatment was defined as at least a 30% reduction from baseline to endpoint (last observation carried forward) in the BPI average pain severity score. BPI is a self-reported scale that measures the severity of pain based on the average pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Response was assessed at endpoint.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 195 | 199
participants | 111 | 97
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in number of patients who achieve a >=30% reduction of the Brief Pain Inventory average pain severity rating after 12 weeks of treatment; Test type: Superiority or Other; p = 0.108, Fisher Exact — p-value is for number of patients who achieve a >=30% reduction of the Brief Pain Inventory average pain severity rating - difference between placebo and duloxetine

5. Secondary Outcome: Number of Responders: 50 Percent (%) or Greater Reduction of the Brief Pain Inventory (BPI) Average Pain Severity Rating at 12 Week Endpoint
Description: Response to treatment was defined as at least a 50% reduction from baseline to endpoint (last observation carried forward) in the BPI average pain severity score. BPI is a self-reported scale that measures the severity of pain based on the average pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Response was assessed at endpoint.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 195 | 199
participants | 95 | 69
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in number of patients who achieve a >=50% reduction of the Brief Pain Inventory average pain severity rating after 12 weeks of treatment; Test type: Superiority or Other; p = 0.006, Fisher Exact — p-value is for number of patients who achieve a >=50% reduction of the Brief Pain Inventory average pain severity rating - difference between placebo and duloxetine

6. Secondary Outcome: Number of Sustained Responders at 12 Week Endpoint
Description: Sustained responders: participants with ≥30% reduction of BPI average pain rating from baseline to endpoint and baseline to earlier visit than last visit and who maintain a ≥20% reduction of BPI average pain rating from baseline at every visit between last visit and earlier visit. BPI: a self-reported scale that measures the severity of pain based on the average pain experienced over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Number of sustained responders was assessed at endpoint.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 195 | 199
participants | 89 | 73
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in number of patients who achieve a >=30% reduction of the Brief Pain Inventory (BPI) average pain severity rating from baseline to endpoint and baseline to earlier visit than last visit and maintains a >=20% reduction of BPI average pain rating from baseline at every visit; Test type: Superiority or Other; p = 0.082, Fisher Exact — p-value is difference between duloxetine and placebo in number of patients who achieve criteria described in null hypothesis

7. Secondary Outcome: Number of Participants Reaching Each Threshold of of BPI Average Pain Score Reduction During the Study - Cumulative Distribution
Description: The results presented are the cumulative number of participants reaching each threshold of BPI average pain reduction. The thresholds are given as percent reductions in BPI average pain score from the baseline score. BPI: a self-reported scale that measures the severity of pain based on the average pain over the past 24-hours. The severity scores range from 0 (no pain) to 10 (pain as severe as you can imagine). Number of participants under each threshold was assessed at endpoint.
Time Frame: 12 weeks
Population: All randomized participants with non-missing baseline value; baseline observation carried forward method was used to impute missing endpoints.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 203 | 198
participants
  Any Increase | 12 | 15
  No Change | 62 | 67
  >0% Decrease | 124 | 121
  >=10% Decrease | 124 | 121
  >=20% Decrease | 116 | 106
  >=30% Decrease | 95 | 83
  >=40% Decrease | 90 | 71
  >=50% Decrease | 85 | 57
  >=60% Decrease | 61 | 38
  >=70% Decrease | 47 | 30
  >=80% Decrease | 32 | 19
  100% Decrease | 15 | 11
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between duloxetine and placebo groups in the empirical cumulated distribution of the percentage pain reduction; Test type: Superiority or Other; p = 0.013, Kolnogorov-Smirnov test — p-value is for difference between duloxetine and placebo groups in the empirical overall cumulated distribution of the percentage pain reduction

8. Secondary Outcome: Change From Baseline to 12 Weeks Endpoint in Clinical Global Impressions of Severity (CGI-S)
Description: Measures severity of illness at the time of assessment compared with start of treatment. Scores range from 1 (normal, not at all ill) to 7 (among the most extremely ill patients). Least Squares Mean values were controlled for investigator and baseline severity.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 195 | 199
units on a scale | -0.95 (0.07) | -0.79 (0.07)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Clinical Global Impression of Severity score after 12 weeks of treatment; Test type: Superiority or Other; p = 0.077, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Clinical Global Impression of Severity score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.16, 95% CI 2-sided [-0.33 to 0.02]

9. Secondary Outcome: Patient's Global Impression of Improvement (PGI-I) at 12 Weeks
Description: A scale that measures the patient's perception of improvement at the time of assessment compared with the start of treatment. The score ranges from 1 (very much better) to 7 (very much worse). Least Squares Mean values were controlled for investigator and baseline severity.
Time Frame: 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 194 | 199
units on a scale | 2.88 (0.09) | 3.19 (0.09)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups Patient's Global Impression of Improvement endpoint value during 12 weeks of treatment; Test type: Superiority or Other; p = 0.011, ANCOVA — p-value is for difference between placebo and duloxetine groups Patient's Global Impression of Improvement endpoint value; Main Effect Model: PGI-I=Treatment+Investigator+Baseline(Type III sums of squares). PGI-Severity score from baseline visit was used as the baseline; Mean Difference (Final Values) = -0.31, 95% CI 2-sided [-0.56 to -0.07]

10. Secondary Outcome: Change From Baseline to 12 Weeks in Roland Morris Disability Questionnaire
Description: Roland-Morris questionnaire will be completed by the patient and measures the degree of disability due to back pain. The questionnaire consists of 24 statements and the patient is instructed to put a mark next to each appropriate statement. The number of statements marked will be added up by the clinician and a total score is given. The total score ranges from 0 (no disability) to 24 (severe disability). Least Squares Mean values were controlled for investigator and baseline severity.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 178 | 179
units on a scale | -2.69 (0.31) | -2.22 (0.32)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Roland Morris Disability Questionnaire total score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.255, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Roland Morris Disability Questionnaire total score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.47, 95% CI 2-sided [-1.28 to 0.34]

11. Secondary Outcome: Change From Baseline to 12 Weeks in Profile of Mood States - Brief Form
Description: The 30-item BPOMS measures mood states and has 6 factors: tension-anxiety (Ten), depression-dejection (Dep), anxiety-hostility (Ang), fatigue (Fat), confusion (Con), and vigor (Vig). Item scores: 0 (not at all) to 4 (extremely). Each factor scores range from 0 to 20. The Total score is sum of all factor scores minus the factor score for vigor (Total=Ten+Dep+Ang+Fat+Con-Vig) and ranges from 0 (least disturbed) to 80 (most disturbed).
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 186 | 188
units on a scale
  Tension-Anxiety - baseline; n=186,n=185 | 4.22 (3.78) | 4.29 (3.70)
  Tension-Anxiety - change; n=186,n=185 | -1.58 (3.48) | -0.78 (3.17)
  Depression-Dejection - baseline; n=185,n=188 | 2.67 (3.63) | 2.74 (3.44)
  Depression-Dejection - change; n=185,n=188 | -0.80 (3.28) | -0.45 (3.07)
  Anger-Hostility - baseline; n=186,n=185 | 2.79 (3.60) | 3.46 (4.11)
  Anger-Hostility - change; n=186,n=185 | -1.18 (3.07) | -0.63 (3.38)
  Vigor-Activity - baseline; n=185, n=187 | 6.77 (4.30) | 7.23 (3.87)
  Vigor-Activity - change; n=185, n=187 | 2.13 (4.53) | 0.81 (3.88)
  Fatigue-Inertia - baseline; n=184, n=188 | 6.49 (4.33) | 6.71 (4.67)
  Fatigue-Inertia - change; n=184, n=188 | -1.74 (3.96) | -1.64 (4.31)
  Confusion-Bewilderment - baseline; n=185, n=187 | 4.09 (2.89) | 4.07 (2.79)
  Confusion-Bewilderment - change; n=185, n=187 | -0.69 (2.71) | -0.14 (2.47)
  Total Mood Disturbance - baseline; n=181, n=180 | 13.31 (16.67) | 14.27 (17.39)
  Total Mood Disturbance - change; n=181, n=180 | -7.90 (14.06) | -4.68 (14.54)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Profile of Mood States Tension-Anxiety subscore during 12 weeks of treatment; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Profile of Mood States Tension-Anxiety subscore; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.88, 95% CI 2-sided [-1.38 to -0.37]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Profile of Mood States Depression-Dejection subscore during 12 weeks of treatment; Test type: Superiority or Other; p = 0.133, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Profile of Mood States Depression-Dejection subscore; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.39, 95% CI 2-sided [-0.90 to 0.12]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Profile of Mood States Anger-Hostility score during 12 weeks of treatment; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Profile of Mood States Anger-Hostility score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.92, 95% CI 2-sided [-1.46 to -0.37]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Profile of Mood States Vigor-Activity score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.003, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Profile of Mood States Vigor-Activity score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 1.13, 95% CI 2-sided [0.38 to 1.88]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Profile of Mood States Fatigue-Inertia score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.469, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Profile of Mood States Fatigue-Inertia score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.25, 95% CI 2-sided [-0.93 to 0.43]
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Profile of Mood States Confusion-Bewilderment score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.006, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Profile of Mood States Confusion-Bewilderment score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -0.57, 95% CI 2-sided [-0.98 to -0.17]
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Profile of Mood States Total Mood Disturbance score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.001, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Profile of Mood States Total Mood Disturbance score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = -4.00, 95% CI 2-sided [-6.41 to -1.60]

12. Secondary Outcome: Change From Baseline to 12 Weeks in 36-item Short-Form (SF-36) Health Survey
Description: The SF-36 Health Status Survey is a generic, health-related scale assessing subjects' quality of life on 8 domains: physical functioning, social functioning, bodily pain, vitality, mental health, role-physical, role-emotional and general health and 2 summary scores (mental component summary [MCS] and physical component summary [PCS]). The score for each of the domain and component summary=0-100 (higher scores indicate better health status or functioning).
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 190 | 188
units on a scale
  Physical Component - baseline; n=147, n=153 | 34.41 (8.18) | 34.29 (7.75)
  Physical Component - change; n=147, n=153 | 6.15 (8.85) | 5.22 (8.25)
  Mental Component - baseline; n=147, n=153 | 49.50 (12.33) | 49.59 (10.35)
  Mental Component - change; n=147, n=153 | 3.34 (9.26) | 0.84 (8.58)
  Bodily Pain - baseline; n=188, n=190 | 33.37 (13.94) | 33.93 (13.81)
  Bodily Pain -change; n=188, n=190 | 18.31 (19.25) | 13.52 (20.15)
  Mental Health - baseline; n=165, n=166 | 69.30 (19.19) | 69.72 (16.73)
  Mental Health - change; n=165, n=166 | 6.65 (15.98) | 1.48 (14.21)
  General Health - baseline; n=188, n=190 | 53.54 (19.31) | 53.11 (22.12)
  General Health - change; n=188, n=190 | 7.81 (17.94) | 5.34 (18.06)
  Physical Functioning - baseline;n=186, n=189 | 50.02 (22.63) | 52.13 (21.17)
  Physical Functioning - change; n=186, n=189 | 13.18 (20.48) | 9.42 (17.63)
  Role-Emotional - baseline; n=172, n=179 | 73.89 (26.63) | 74.21 (25.64)
  Role-Emotional - change; n=172, n=179 | 8.19 (21.90) | 5.12 (23.52)
  Role-Physical - baseline; n=172, n=179 | 46.77 (22.37) | 46.42 (23.68)
  Role-Physical - change; n=172, n=179 | 12.97 (22.24) | 11.66 (22.89)
  Social Functioning -baseline; n=188, n=190 | 67.02 (24.28) | 69.67 (24.03)
  Social Functioning - change; n=188, n=190 | 12.70 (22.18) | 7.11 (21.02)
  Vitality - baseline; n=163, n=165 | 50.69 (19.08) | 48.64 (18.92)
  Vitality - change; n=163, n=165 | 9.33 (18.94) | 6.30 (18.40)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the 36-SF Health Survey Physical Component score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.168, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the 36-SF Health Survey Physical Component score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 1.24, 95% CI 2-sided [-0.53 to 3.02]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the SF-36 Health Survey Mental Component score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.010, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the SF-36 Health Survey Mental Component score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 2.24, 95% CI 2-sided [0.53 to 3.96]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the SF-36 Health Survey Bodily Pain Transformed score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.016, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the SF-36 Health Survey Bodily Pain Transformed score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 4.58, 95% CI 2-sided [0.86 to 8.30]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the SF-36 Health Survey Mental Health Transformed score during 12 weeks of treatment; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the SF-36 Health Survey Mental Health Transformed score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 4.88, 95% CI 2-sided [2.15 to 7.61]
Statistical Analysis 5: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the SF-36 Health Survey General Health Transformed score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.101, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the SF-36 Health Survey General Health Transformed score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 2.58, 95% CI 2-sided [-0.50 to 5.67]
Statistical Analysis 6: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the SF-36 Health Survey Physical Functioning Transformed score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.058, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the SF-36 Health Survey Physical Functioning Transformed score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 3.50, 95% CI 2-sided [-0.12 to 7.12]
Statistical Analysis 7: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the SF-36 Health Survey Role-Emotional Transformed score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.227, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the SF-36 Health Survey Role-Emotional Transformed score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 2.43, 95% CI 2-sided [-1.52 to 6.37]
Statistical Analysis 8: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the SF-36 Health Survey Role-Physical Transformed score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.383, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the SF-36 Health Survey Role-Physical Transformed score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 1.91, 95% CI 2-sided [-2.39 to 6.21]
Statistical Analysis 9: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the SF-36 Health Survey Social Functioning Transformed score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.030, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the SF-36 Health Survey Social Functioning Transformed score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 4.00, 95% CI 2-sided [0.38 to 7.61]
Statistical Analysis 10: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the SF-36 Health Survey Vitality Transformed score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.022, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the SF-36 Health Survey Vitality Transformed score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 4.10, 95% CI 2-sided [0.59 to 7.60]

13. Secondary Outcome: Change From Baseline to 12 Weeks in European Quality of Life Questionnaire - 5 Dimension
Description: Generic, multidimensional, health-related, quality-of-life instrument. The profile allows patients to rate their health state in 5 health domains: mobility, self-care, usual activities, pain/discomfort, and mood. A single score between 1 and 3 is generated for each domain. For each patient, the outcome rating on 5 domains will be mapped to a single index through an algorithm. The index ranges between 0 and 1; higher scores indicate a better health state perceived by the patient. Participants were evaluated with the United Kingdom (UK) and the United States (US) population based index score.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 190 | 192
units on a scale
  UK population-based Index Score-baseline | 0.52 (0.27) | 0.57 (0.24)
  UK population-based Index Score-change | 0.19 (0.31) | 0.07 (0.26)
  US population-based Index Score-baseline | 0.66 (0.17) | 0.69 (0.16)
  US population-based Index Score-change | 0.12 (0.21) | 0.05 (0.17)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the European Quality of Life Questionnaire - 5 Dimension - United Kingdom population-based Index score during 12 weeks of treatment; Test type: Superiority or Other; p < 0.001, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the European Quality of Life Questionnaire - 5 Dimension - United Kingdom population-based Index score; Main Effect Model: Change = Treatment + Investigator (Type III sums of squares); Mean Difference (Final Values) = 0.07, 95% CI 2-sided [0.03 to 0.12]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the European Quality of Life Questionnaire - 5 Dimension - United States population-based index score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.002, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the European Quality of Life Questionnaire - 5 Dimension - United States population-based index score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 0.05, 95% CI 2-sided [0.02 to 0.08]

14. Secondary Outcome: Change From Baseline to 12 Weeks in Work Productivity and Activity Impairment Instrument (WPAI)
Description: WPAI: self-administered instrument used to measure effect of general health and symptom severity on work productivity and regular activities and yields 4 types of scores: Absenteeism (work time missed); Presenteeism (impairment at work/reduced on-the-job effectiveness); Work Productivity Loss (overall work impairment/absenteeism plus presenteeism); and Activity Impairment.
  1. Absenteeism
  2. Presenteeism
  3. Work productivity loss
  4. Activity Impairment Scores range from 0 to 1 for each of the above 4 types; higher scores indicate greater impairment.
Time Frame: baseline, 12 weeks
Population: All randomized participants with baseline and at least 1 non-missing post-baseline value. Last observation carried forward method was used to impute missing endpoints. Not for all participants were data for all WPAI items available.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 190 | 196
units on a scale
  Absenteeism, baseline; n=79, n=93 | 0.08 (0.20) | 0.10 (0.25)
  Absenteeism, change; n=79, n=93 | -0.03 (0.18) | -0.03 (0.18)
  Presenteeism, baseline; n=79, n=90 | 0.49 (0.25) | 0.48 (0.22)
  Presenteeism, change; n=79, n=90 | -0.22 (0.24) | -0.18 (0.23)
  Work Productivity Loss, baseline; n=77, n=89 | 0.50 (0.25) | 0.50 (0.23)
  Work Productivity Loss, change; n=77, n=89 | -0.22 (0.26) | -0.18 (0.25)
  Activity Impairment, baseline; n=190, n=196 | 0.56 (0.22) | 0.56 (0.19)
  Activity Impairment, change; n=190, n=196 | -0.23 (0.25) | -0.17 (0.21)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Work Productivity and Activity Impairment Instrument (WPAI) - Absenteeism score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.461, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Work Productivity and Activity Impairment Instrument (WPAI) - Absenteeism score; Main Effect Model: Change = Treatment + Investigator + Baseline (Type III sums of squares); Mean Difference (Final Values) = 0.02, 95% CI 2-sided [-0.03 to 0.06]
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Work Productivity and Activity Impairment Instrument (WPAI) - Presenteeism score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.374, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Work Productivity and Activity Impairment Instrument (WPAI) - Presenteeism score; Mean Difference (Final Values) = -0.03, 95% CI 2-sided [-0.09 to 0.03]
Statistical Analysis 3: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Work Productivity and Activity Impairment Instrument (WPAI) - Work Productivity Loss score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.557, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Work Productivity and Activity Impairment Instrument (WPAI) - Work Productivity Loss score; Mean Difference (Final Values) = -0.02, 95% CI 2-sided [-0.09 to 0.05]
Statistical Analysis 4: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of the Work Productivity and Activity Impairment Instrument (WPAI) - Activity Impairment score during 12 weeks of treatment; Test type: Superiority or Other; p = 0.007, ANCOVA — p-value is for difference between placebo and duloxetine groups in change of the Work Productivity and Activity Impairment Instrument (WPAI) - Activity Impairment score; Mean Difference (Final Values) = -0.06, 95% CI 2-sided [-0.10 to -0.02]

15. Secondary Outcome: Participants Who Discontinued From Baseline to 12 Weeks
Description: Reasons for discontinuation are listed in the participant flow.
Time Frame: baseline, 12 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 198 | 203
participants | 51 | 47

16. Secondary Outcome: Change From Baseline to 12 Weeks in Uric Acid
Description: Least Squares Mean values were controlled for investigator.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Micromole/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 190 | 194
Micromole/Liter | -14.06 (4.60) | 1.34 (4.64)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of uric acid during 12 weeks of treatment; Test type: Superiority or Other; p = 0.010, ANOVA — p-value is for difference between placebo and duloxetine groups in uric acid - change; Change Variable = Treatment + Investigator (Type III sums of squares). Rank-transformed change was used as change variable in the ANOVA model

17. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Albumin
Description: Least Squares Mean values were controlled for investigator.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Deviation); unit: Gram/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 190 | 194
Gram/Liter | -0.76 (0.23) | -0.12 (0.23)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of Albumin during 12 weeks of treatment; Test type: Superiority or Other; p = 0.031, ANOVA — p-value is for difference between duloxetine and placebo in albumin - change

18. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Alkaline Phosphatase
Description: Least Squares Mean values were controlled for investigator.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 190 | 194
Units/Liter | 1.59 (0.94) | -1.85 (0.94)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of alkaline phosphatase during 12 weeks of treatment; Test type: Superiority or Other; p = 0.004, ANOVA — p-value is for difference between duloxetine and placebo in alkaline phosphatase - change

19. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Alanine Aminotransferase
Description: Least Squares Mean values were controlled for investigator.
Time Frame: baseline, 12 weeks
Population: All randomized participants with baseline and at least 1 non-missing post-baseline value. Last observation carried forward method was used to impute missing.
  endpoints.
Measure: Least Squares Mean (Standard Error); unit: Units/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 190 | 194
Units/Liter | 1.51 (1.01) | -1.71 (1.01)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of Alanine Aminotransferase during 12 weeks of treatment; Test type: Superiority or Other; p = 0.013, ANOVA — p-value is for difference between duloxetine and placebo in alanine aminotransferase - change

20. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Aspartate Aminotransferase
Description: Least Squares Mean values were controlled for investigator.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Units/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 190 | 194
Units/Liter | 1.90 (0.92) | -0.54 (0.92)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of aspartate aminotransferase during 12 weeks of treatment; Test type: Superiority or Other; p = 0.039, ANOVA — p-value for difference between duloxetine and placebo in aspartate aminotransferase - change

21. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Creatinine
Description: Least Squares Mean values were controlled for investigator.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Micromole/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 190 | 194
Micromole/Liter | -1.69 (0.82) | 0.70 (0.82)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of creatinine during 12 weeks of treatment; Test type: Superiority or Other; p = 0.024, ANOVA — p-value is for difference between duloxetine and placebo in creatinine - change

22. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Total Protein
Description: Least Squares Mean values were controlled for investigator.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: Gram/Liter
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 190 | 194
Gram/Liter | -1.34 (0.30) | -0.43 (0.30)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of total protein during 12 weeks of treatment; Test type: Superiority or Other; p = 0.019, ANOVA — p-value is for difference between duloxetine and placebo in total protein - change

23. Secondary Outcome: Change From Baseline to 12 Weeks in Blood Pressure
Description: Least Squares Mean values were controlled for investigator.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: millimeter mercury
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 194 | 198
millimeter mercury
  Systolic Blood Pressure (millimeter mercury) | 0.49 (0.85) | -0.59 (0.85)
  Diastolic Blood Pressure (millimeter mercury) | -0.14 (0.67) | -0.64 (0.67)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of systolic blood pressure during 12 weeks of treatment; Test type: Superiority or Other; p = 0.329, ANOVA — p-value is for difference between placebo and duloxetine groups in change of systolic blood pressure; Main Effect Model: Change = Treatment + Investigator (Type III sums of squares)
Statistical Analysis 2: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of diastolic blood pressure during 12 weeks of treatment; Test type: Superiority or Other; p = 0.562, ANOVA — p-value is for difference between placebo and duloxetine groups in change of diastolic blood pressure; Main Effect Model: Change = Treatment + Investigator (Type III sums of squares)

24. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Weight
Description: Least Squares Mean values were controlled for investigator.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: kilogram
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 194 | 198
kilogram | -0.31 (0.17) | 0.05 (0.17)

25. Secondary Outcome: Change From Baseline to 12 Week Endpoint in Pulse Rate
Description: Least Squares Mean values were controlled for investigator.
Time Frame: baseline, 12 weeks
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: beats per minute
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 194 | 198
beats per minute | 0.18 (0.65) | -0.17 (0.64)
Statistical Analysis 1: Comparison: Duloxetine vs Placebo; Tested was the null hypothesis that there is no difference between placebo and duloxetine groups in change of pulse rate during 12 weeks of treatment; Test type: Superiority or Other; p = 0.680, ANOVA — p-value is for difference between duloxetine and placebo in pulse rate - change

26. Secondary Outcome: Number of Participants With Suicidal Ideation or Suicidal Behaviors According to the Columbia Suicide Severity Rating Scale
Description: The Columbia Suicide Severity Rating Scale (C-SSRS) captures the occurrence, severity, and frequency of suicide-related thoughts and behaviors during the assessment period. The scale includes suggested questions to solicit the type of information needed to determine if a suicide-related thought or behavior occurred.
Time Frame: baseline through 12 weeks
Population: All randomized participants.
Measure: Number; unit: participants
Arm/Group | Duloxetine | Placebo
Number analyzed (Participants) | 198 | 203
participants | 0 | 0

ADVERSE EVENTS:
Arm/Group | Duloxetine | Placebo
Serious Adverse Events (participants affected / at risk) | 5/198 | 0/203
Other Adverse Events (participants affected / at risk) | 123/198 | 112/203
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=198) | Placebo (N=203)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0)
Alcohol poisoning (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Myopathy toxic (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0)
Asthma (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Duloxetine (N=198) | Placebo (N=203)
Tachycardia (Cardiac disorders) | 0 (0) | 3 (3)
Tinnitus (Ear and labyrinth disorders) | 2 (2) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 5 (5) | 3 (3)
Vision blurred (Eye disorders) | 2 (2) | 1 (1)
Abdominal pain upper (Gastrointestinal disorders) | 2 (2) | 4 (5)
Constipation (Gastrointestinal disorders) | 12 (12) | 7 (7)
Diarrhoea (Gastrointestinal disorders) | 9 (9) | 6 (6)
Dry mouth (Gastrointestinal disorders) | 13 (14) | 4 (4)
Flatulence (Gastrointestinal disorders) | 3 (3) | 2 (2)
Nausea (Gastrointestinal disorders) | 35 (35) | 6 (7)
Toothache (Gastrointestinal disorders) | 2 (2) | 0 (0)
Vomiting (Gastrointestinal disorders) | 3 (3) | 3 (3)
Asthenia (General disorders) | 2 (2) | 0 (0)
Fatigue (General disorders) | 7 (7) | 3 (3)
Hypertransaminasaemia (Hepatobiliary disorders) | 2 (2) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 4 (4)
Influenza (Infections and infestations) | 3 (4) | 5 (5)
Nasopharyngitis (Infections and infestations) | 5 (5) | 4 (4)
Respiratory tract infection viral (Infections and infestations) | 0 (0) | 3 (3)
Rhinitis (Infections and infestations) | 2 (2) | 2 (2)
Sinusitis (Infections and infestations) | 1 (1) | 3 (3)
Upper respiratory tract infection (Infections and infestations) | 4 (5) | 8 (9)
Viral infection (Infections and infestations) | 2 (2) | 0 (0)
Joint sprain (Injury, poisoning and procedural complications) | 2 (2) | 0 (0)
Blood creatine phosphokinase increased (Investigations) | 0 (0) | 3 (3)
Anorexia (Metabolism and nutrition disorders) | 4 (4) | 0 (0)
Decreased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Hypertriglyceridaemia (Metabolism and nutrition disorders) | 0 (0) | 3 (3)
Increased appetite (Metabolism and nutrition disorders) | 2 (2) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 (1) | 7 (9)
Back pain (Musculoskeletal and connective tissue disorders) | 3 (3) | 3 (3)
Muscle spasms (Musculoskeletal and connective tissue disorders) | 2 (2) | 0 (0)
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 (2) | 4 (4)
Neck pain (Musculoskeletal and connective tissue disorders) | 2 (4) | 1 (1)
Dizziness (Nervous system disorders) | 10 (10) | 3 (3)
Headache (Nervous system disorders) | 27 (54) | 25 (35)
Migraine (Nervous system disorders) | 2 (2) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 3 (3)
Somnolence (Nervous system disorders) | 10 (10) | 2 (2)
Tension headache (Nervous system disorders) | 0 (0) | 3 (3)
Anxiety (Psychiatric disorders) | 2 (2) | 2 (2)
Confusional state (Psychiatric disorders) | 2 (2) | 0 (0)
Insomnia (Psychiatric disorders) | 5 (5) | 6 (6)
Libido decreased (Psychiatric disorders) | 4 (4) | 1 (1)
Urinary retention (Renal and urinary disorders) | 2 (2) | 0 (0)
Urine flow decreased (Renal and urinary disorders) | 2 (2) | 0 (0)
Ejaculation disorder (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Sexual dysfunction (Reproductive system and breast disorders) | 2 (2) | 0 (0)
Yawning (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 0 (0)
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 5 (5) | 2 (2)
Pruritus (Skin and subcutaneous tissue disorders) | 2 (3) | 1 (1)
Hypertension (Vascular disorders) | 2 (2) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days